CLINICAL TRIAL: NCT05484076
Title: The Effect of Lactation Counseling on Breastfeeding Behaviors of Women: A Randomized Controlled Longitudinal Study
Brief Title: The Effect of Lactation Counseling on Breastfeeding Behaviors of Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Tugce Sonmez, Principal Investigator, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 200720asel
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Breastfeeding; Mothers
Keywords: baby; breastfeeding; counseling; mother; telehealth
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- breastfeeding counseling (Experimental): Pregnant women will be given breastfeeding counseling, which will take place in a total of five sessions at specified intervals.
  Interventions: Other: breastfeeding counseling
- control group (No Intervention): No training will be given to the control group. They will be asked to fill in the questionnaires included in our study at specified intervals.

INTERVENTIONS:
Other: breastfeeding counseling — A breastfeeding booklet will be created by the researchers by taking expert opinion. This booklet will explain everything about breastfeeding in five sessions.
  At 34-38 weeks of pregnancy, the first interviews will be done face-to-face at the hospital. The second interview will be made face-to-face or online, depending on the conditions, in the first 1-5 days after the birth. Subsequent interviews (postpartum 1-4 weeks, postpartum 5-12 weeks, postpartum 13-24 weeks) will be held online. The scales used in the research will be applied twice, before and after the training.
  Arms: breastfeeding counseling

SUMMARY:
Breast milk is the main source of nutrition for newborns. Although breastfeeding is seen as a necessary process to meet the nutritional needs of babies in the early stages of life, it has a key role for a healthy generation in the long run. In this respect, the article has a unique value for a sustainable future in terms of its effects on the mother and baby in particular and on the social level in general. The study was planned as a randomized controlled longitudinal study. The research is planned to be carried out between September 2022 and January 2023 in Çukurova University Medical Faculty Balcalı Training and Research Hospital pregnant outpatient clinic. The sample of the study will consist of 104 pregnant women, 52 of whom are in the experimental group and 52 in the control group, determined by power analysis. A training module will be created by taking expert opinions. The training module will consist of 5 sessions. Each session will last 1 hour, with 45 minutes of interactive lecture and 15 minutes of question and answer. Module sessions will have a dynamic structure that takes into account the needs of mother and baby during pregnancy and postpartum period. At 34-38 weeks of pregnancy, the first interviews are face-to-face at the hospital, the second interview is postpartum 1-5. day depending on the conditions, face-to-face or online, subsequent meetings will be held online. During the implementation phase, quantitative measurements of the research will be carried out by using the "Antenatal Pregnant Information Form", "Postnatal Mother Information Form", " The Infant Breastfeeding Assesment Tool", "Breastfeeding Motivation Scale", IOWA Infant Nutrition Attitude Scale" and " Mother-To-İnfant Bonding Scale".

DETAILED DESCRIPTION:
Breast milk is the main source of nutrition for newborns. Although breastfeeding is seen as a necessary process to meet the nutritional needs of babies in the early stages of life, it has a key role for a healthy generation in the long run. In this respect, the project has a unique value for a sustainable future in terms of its effects on the mother and baby in particular and on the social level in general. It is basically a human right that every baby has the potential for a healthy future by being fed with breast milk. In particular, the disruptions experienced in health services during the pandemic process have also significantly affected maternal and child health services. In this respect, another unique value is that it is a longitudinal study that includes innovative methods to be taken at the national level to quickly compensate for the lost momentum in breastfeeding during the pandemic process. Face-to-face counseling and training will start during pregnancy, and then continue as telehealth services. Continuity of counseling will increase the mother's compliance with breastfeeding. Behavior change, which will be developed individually, will also positively affect mother-infant harmony and family-spouse harmony, thus supporting the creation of a healthy development environment. Another unique value of the study is that it will provide data on the comparison of innovative education methods with traditional education methods. Thus the findings obtained will help to improve, regulate or build capacity of future initiatives.

The study was planned as a randomized controlled longitudinal study. The research is planned to be carried out between September 2022 and January 2023 in Çukurova University Medical Faculty Balcalı Training and Research Hospital pregnant outpatient clinic. The sample of the study will consist of 104 pregnant women, 52 of whom are in the experimental group and 52 in the control group, determined by power analysis. A training module will be created by taking expert opinions. The training module will consist of 5 sessions. Each session will last 1 hour, with 45 minutes of interactive lecture and 15 minutes of question and answer. Module sessions will have a dynamic structure that takes into account the needs of mother and baby during pregnancy and postpartum period. At 34-38 weeks of pregnancy, the first interviews are face-to-face at the hospital, the second interview is postpartum 1-5. day depending on the conditions, face-to-face or online, subsequent meetings will be held online. During the implementation phase, quantitative measurements of the research will be carried out by using the "Antenatal Pregnant Information Form", "Postnatal Mother Information Form", " The Infant Breastfeeding Assesment Tool", "Breastfeeding Motivation Scale", IOWA Infant Nutrition Attitude Scale" and " Mother-To-İnfant Bonding Scale".

the scope of the widespread effect of our research; The training booklet prepared with the expert opinion for the training process will be brought to the field.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Not having received breastfeeding counseling before
* Being her first pregnancy
* Those who have a communication device that can use and download Teknolojik-Online systems (Smartphone, message, Google forms, zoom, whatsaap)
* Not having a vision-hearing problem
* Ability to read and write
* Last trimester (34 and above gestational weeks)
* Single pregnancy
* Giving birth at term (38-40 weeks)
* The newborn does not have health problems that require hospitalization

Exclusion Criteria:

* Maternal (mastectomy, breast-milk infection and drug use, psychiatric diseases, etc.) preventing breastfeeding,
* Fetal (cleft palate, chromosomal anomalies, neurological diseases that may adversely affect breastfeeding, etc.)
* Unwillingness to continue research
* Having situations that require separation of mother and baby in the postpartum period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-10-29 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Antenatal Pregnant Information Form | 34-38 weeks of pregnancy
  This form, which was prepared by the researchers in line with the literature, consists of 11 questions containing the sociodemographic characteristics of pregnant women and pregnancy information.
Postnatal Mother Information Form | postpartum 1-5 day
  this form, which was prepared in line with the literature review, consists of 18 questions that include information on mothers regarding the postpartum period, breastfeeding and baby.
The Infant Breastfeeding Assesment Tool | postpartum first 6 months
  The scale is a measurement tool developed to determine temporary feeding difficulties in the first 4 to 5 days in healthy and term babies. The scale consists of six questions and the evaluation is made by the mothers. Scoring is done on the basis of the mothers' answers to the questions. Each question is evaluated between 0-3 points (min:0, max:12). Getting a high score from the scale means that there is better. If the baby carries all the effective feeding behaviors, the grand total is 12 points. The score range for effectively fed infants is 10-12 points. The score range for babies who breastfeed quite successfully when encouraged is 7-9 points, and feeding is considered moderately effective. Babies who do not start feeding with stimuli, do not seek or breastfeed for short periods are evaluated in the range of 0-6 points. With this tool, maternal satisfaction and comfort during breastfeeding can also be evaluated.
Breastfeeding Motivation Scale | postpartum first 6 months
  For multiparous mothers, it was determined by explanatory factor analysis that it consisted of 24 items and six sub-factors. According to the calculated Cronbach's alpha value, the Breastfeeding Motivation Scale is a very reliable scale for primiparous (cronbach's alpha: 0.887) and multiparous (cronbach's alpha: 0.914) mothers. The scale consists of 24 items and 5 sub-dimensions. The scale items are in 4-point Likert type, and each item is scored between 1-4 (min:24, max:96).The score of the sub-dimensions is calculated by taking the total score of the scale and the average of the sub-dimension scores of the scale. As the score obtained from the scale sub-dimension increases, it is interpreted as an increase in the motivation representing that sub-dimension. As the score obtained from the scale sub-dimension increases, it is interpreted as an increase in the motivation representing that sub-dimension.
Iowa Infant Nutrition Attitude Scale | postpartum first 6 months
  The scale was developed in order to evaluate women's attitudes towards breastfeeding and to evaluate the duration of breastfeeding together with the choice of baby feeding method. The scale consists of 17 questions and the answers range from 1 (strongly disagree) to 5 (strongly agree). While 9 questions in the scale support breastfeeding, 8 items contain a supportive approach to formula feeding. The total score that can be obtained from the scale is between min: 17 and max: 85.
  Total scale scores can be further categorized into groups:
  1. positive to breastfeeding (scale score 70-85),
  2. neutral (IIFAS score 49-69), and
  3. positive to formula feeding (scale score 17-48).
Mother-To-İnfant Bonding Scale | postpartum first 6 months
  In 2005, Taylor et al. The scale developed by Karakulak and Alparslan was adapted to Turkish. The scale, which allows the mother to describe her feelings towards her baby with a single word, can be applied from the first day after birth. It reveals the relationship between the bond established and the mother's first period mood. The scale is in a 4-point Likert format, consisting of 8 items. The answers consisting of four options are scored between 0-3. The scale min:0, max: 24 score. In the evaluation, the 1st, 4th, and 6th items are positive emotion expressions and are scored as 0,1,2,3; 2.,3.,5.,7. Items 8 and 8 are negative emotional expressions and are scored as 3,2,1,0 and reversely. It has been reported that the inter-rater reliability of the scale is 0.71 and the Cronbach's Alpha is 0.66. High scale scores are interpreted as an increase in mother-infant attachment.

CONTACTS AND LOCATIONS:
Overall Officials: tuğçe sönmez, PhD, Principal Investigator — Tarsus University
Locations (1):
- Tuğçe Sönmez, Toroslar, Mersin, Turkey (Türkiye)

REFERENCES:
- [Derived] Sonmez T, Surucu SG, Vurgec BA. Effects of hybrid breastfeeding counseling on women's breastfeeding behaviors: a randomized controlled longitudinal study. BMC Pregnancy Childbirth. 2025 Jun 7;25(1):663. doi: 10.1186/s12884-025-07781-z. PMID 40483454